CLINICAL TRIAL: NCT01250236
Title: Effect of Brimonidine on Corneal Thickness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Augenarztpraxis Breisach (Other)
Responsible Party: PD Dr. Matthias Grueb, Augenarztpraxis Breisach
Other Study IDs: Grueb Klin CT
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Impact of Brimonidine on the Cornea
Keywords: brimonidine; alpha-2 adrenoceptor; cornea; corneal thickness
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- verum: brimonidine 0.1% eye drops twice daily
  Interventions: Drug: brimonidine 0.1%
- placebo: sodium hyaluronate 1.8mg/ml eye drops twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: brimonidine 0.1% — brimonidine 0.1% eye drops twice daily
  Groups: verum
Drug: placebo — sodium hyaluronate 1.8mg/ml eye drops twice daily
  Groups: placebo

SUMMARY:
Brimonidine, an alpha-2 adrenoceptor agonist, is an effective and safe medication which is widely used in glaucoma treatment. Although it is known that it is quickly taken up by the cornea following topical administration and that the cornea has alpha-2 adrenoceptors there are only few studies available on the impact brimonidine has on the cornea. The aim of the study is to find out

1. whether topical administration of brimonidine results in interaction with corneal alpha-2 adrenoceptors in terms of an increase in corneal thickness and
2. whether there are any differences between the response corneal epithelium, stroma and endothelium show to alpha-2 adrenoceptor stimulation.

ELIGIBILITY:
Inclusion Criteria:

* healthy, 18-99 years, normal ophthalmologic history, consent to participate in the study

Exclusion Criteria:

* any serious medical or neurologic conditions and/or regular use of local or systemic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: consecutive
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
corneal thickness | 5 days

SECONDARY OUTCOMES:
intraocular pressure | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Grueb, Priv. Doz. Dr., Study Director — Augenarztpraxis Breisach
Locations (1):
- Augenarztpraxis, Breisach, Baden-Wurttemberg, Germany